CLINICAL TRIAL: NCT07317960
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Trial to Evaluate the Safety and Tolerability of PollenVax, a Subcutaneous Emulsion, in Patients With Mugwort Pollen-Induced Allergic Rhinitis
Brief Title: Phase I Study of PollenVax in Patients With Mugwort Pollen-Induced Allergic Rhinitis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kazakh National Agrarian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POL-I-30-2025; BR25293305 (Other Grant/Funding Number: The Ministry of Health of the Republic of Kazakhstan)
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Allergic Rhinitis Due to Artemisia Pollen
Keywords: Mugwort Pollen Allergy; Artemisia Allergy; Allergen-Specific Immunotherapy; recombinant Artemisia pollen major allergen Art v 1; an ultra-short subcutaneous allergen-specific immunotherapy regimen

STUDY DESIGN:
Intervention Model Description: Participants are randomized in parallel to receive either the investigational product (PollenVax) or placebo and remain in their assigned treatment group throughout the study without crossover.
Who Masked: Participant, Care Provider, Investigator
Masking Description: No additional parties are masked beyond those listed above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PollenVax (Experimental): Participants receive PollenVax, a recombinant allergen-based vaccine containing recombinant Artemisia pollen major allergen Art v 1 formulated with Montanide ISA 51 adjuvant, administered subcutaneously in an ultra-short immunotherapy regimen.
  Interventions: Biological: PollenVax
- Placebo Comparator (Placebo Comparator): Participants receive a matching placebo emulsion for subcutaneous administration according to the same schedule as the investigational product.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PollenVax — PollenVax is a recombinant allergen-based vaccine containing recombinant Artemisia pollen major allergen Art v 1 formulated with Montanide ISA 51 adjuvant. The vaccine is administered subcutaneously in an ultra-short allergen-specific immunotherapy regimen consisting of four injections.
  Arms: PollenVax
Other: Placebo — The placebo is a matching emulsion for subcutaneous administration without the active recombinant allergen, administered according to the same schedule as the investigational product.
  Arms: Placebo Comparator

SUMMARY:
This Phase I randomized, double-blind, placebo-controlled clinical trial evaluates the safety and tolerability of PollenVax, a novel recombinant allergen-based vaccine for allergen-specific immunotherapy, in adult patients with mugwort pollen-induced allergic rhinitis.

DETAILED DESCRIPTION:
This single-center Phase I randomized, double-blind, placebo-controlled study is designed to assess the safety, tolerability, and immunogenicity of PollenVax, a recombinant allergen-based vaccine containing Artemisia pollen major allergen Art v 1 formulated with Montanide ISA 51 adjuvant.

The study evaluates an ultra-short subcutaneous allergen-specific immunotherapy regimen consisting of four weekly injections administered during the remission period outside the active pollen season.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent, dated and signed by the participant and the investigator prior to any study-related procedures;
2. Male or female participants;
3. Age 18 to 65 years, inclusive;
4. Ability and willingness to comply with all study procedures and attend all scheduled study visits for medical follow-up;
5. Patients with allergic rhinitis as the primary diagnosis, of moderate to severe severity, caused by mugwort pollen (Artemisia vulgaris) for at least two years, in accordance with the recommendations of Allergic Rhinitis and its Impact on Asthma (ARIA); patients may have well-controlled asthma as a comorbid condition, of mild to moderate severity, according to the Global Initiative for Asthma (GINA 2022-2024) guidelines, or no asthma;
6. A positive skin prick test to Artemisia vulgaris with a wheal diameter of ≥ 3 mm, confirmed using appropriate positive and negative controls;
7. Presence of specific immunoglobulin E (IgE) to Artemisia vulgaris major allergen Art v 1 at Class ≥ 2, determined using ImmunoCAP technology;
8. Sensitization to Artemisia vulgaris associated with clinically significant allergic symptoms for which allergen-specific immunotherapy (ASIT) is indicated;
9. Laboratory and instrumental test results within normal ranges or showing deviations not considered clinically significant by the investigator;
10. Body mass index (BMI) between 18.5 and 30.0 kg/m², inclusive;
11. Normal body temperature, defined as 35.5 °C to 36.6 °C, inclusive;
12. Resting blood pressure within the following ranges:

    * Systolic blood pressure (SBP): 120-129 mmHg
    * Diastolic blood pressure (DBP): 60-89 mmHg
13. For women of childbearing potential, a negative pregnancy test at screening;
14. Agreement to use adequate contraception methods from screening until 90 days after completion of the study.

Exclusion Criteria:

1. Previous allergen-specific immunotherapy (ASIT) to Artemisia vulgaris or any other cross-reactive allergen within the past 5 years, or current ASIT to any allergen;
2. Concomitant sensitization that may interfere with study conduct or interpretation, particularly if the skin prick test response to another allergen exceeds that to Artemisia vulgaris;
3. Severe asthma or forced expiratory volume in 1 second (FEV₁) ≤ 80% predicted, even if pharmacologically controlled;
4. History of severe systemic reactions to allergen-specific immunotherapy;
5. Complications of allergic rhinitis at screening, including allergic sinusitis, nasal polyps, tonsillitis, or otitis media;
6. Treatment with immunoglobulin therapy;
7. Completed or ongoing treatment with anti-IgE monoclonal antibodies (e.g., omalizumab) and/or immune checkpoint inhibitors;
8. Immune system disorders, including autoimmune diseases or immunodeficiency states, except for well-controlled Hashimoto's thyroiditis or type 1 diabetes mellitus;
9. Severe acute or chronic inflammatory or infectious diseases;
10. Decompensated comorbid conditions, including severe, unstable, or uncontrolled somatic diseases based on medical history, such as:

    1. Severe respiratory failure;
    2. Liver cirrhosis Child-Pugh class B or C;
    3. Severe or unstable angina pectoris;
    4. Chronic heart failure NYHA class III-IV or decompensated heart failure;
    5. Uncontrolled arterial hypertension (systolic blood pressure >130 mmHg and/or diastolic blood pressure >90 mmHg);
    6. Uncontrolled cardiac arrhythmias, including Lown class IVb or V ventricular arrhythmias or bifascicular intraventricular block;
    7. Myocardial infarction, acute cerebrovascular accident, transient ischemic attack, or pulmonary embolism within 6 months prior to study entry (Visit 0), or large aortic aneurysm (>6 cm);
    8. Coronary artery bypass grafting or coronary stenting within 3 months prior to study entry (Visit 0);
    9. Any other condition that, in the opinion of the investigator, may interfere with interpretation of study results or limit the participant's ability to complete the study;
    10. Malignancy of any localization currently or within 5 years prior to enrollment, except for completely treated carcinoma in situ;
    11. History of severe renal insufficiency;
    12. History of severe hepatic insufficiency;
    13. Human immunodeficiency virus (HIV) infection, syphilis, hepatitis B virus, and/or hepatitis C virus infection;
11. Exacerbation of chronic allergic skin diseases (e.g., atopic dermatitis, generalized urticaria) as determined by physical examination;
12. Substance abuse, including alcohol, narcotics, or prescription drug abuse, within the past year and/or during the study;
13. For women of reproductive potential: pregnancy and/or lactation;
14. For women: unprotected sexual intercourse with a non-sterilized male partner within 30 days prior to screening;
15. Systemic or local (including ophthalmic) beta-blocker therapy;
16. Use of prohibited medications, including but not limited to:

    * Systemic leukotriene receptor antagonists (e.g., montelukast);
    * Systemic ketotifen;
    * Beta-blockers (systemic or topical);
    * Medications containing terfenadine, theophylline or its derivatives;
    * Roflumilast or other phosphodiesterase-4 (PDE-4) inhibitors;
    * Pseudoephedrine, tiotropium, or other anticholinergic agents;
    * Cromones or mast cell stabilizers;
    * Phenothiazines;
    * Immunosuppressive therapy;
    * Antiviral or antibacterial vaccination within 14 days before and 7 days after administration of the investigational product;
17. Contraindications to epinephrine administration, including but not limited to symptomatic ischemic heart disease, severe hypertension, hyperthyroidism, or glaucoma;
18. Severe psychiatric or neurological disorders, or completed or ongoing long-term treatment with tranquilizers or psychoactive medications, including tricyclic antidepressants;
19. Legally incapacitated individuals;
20. Participants considered to be at high risk of non-compliance with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of PollenVax after four subcutaneous administrations | From first administration through 50 days after the last injection
  Evaluation of the safety and tolerability of PollenVax based on the incidence, severity, and relationship to study treatment of adverse events (AEs) and serious adverse events (SAEs) following four subcutaneous administrations in patients with mugwort pollen-induced seasonal allergic rhinitis during the remission period outside the active pollen season.
Frequency and pattern of adverse events following administration of PollenVax | From first administration through 50 days after the last injection
  Assessment of the frequency, type, and severity of local and systemic adverse events occurring after four subcutaneous administrations of PollenVax, including identification of the most commonly observed adverse events.

SECONDARY OUTCOMES:
Dose-related safety profile of PollenVax | From first administration through 50 days after the last injection
  Evaluation of the relationship between administered dose levels of PollenVax and the occurrence and severity of adverse events in patients with mugwort pollen-induced seasonal allergic rhinitis.
Humoral immunogenicity of PollenVax | Baseline to Day 50
  Assessment of humoral allergen-specific immune response based on changes in serum levels of allergen-specific IgE and IgG4 antibodies to Artemisia pollen major allergen Art v 1 measured before and after allergen-specific immunotherapy.
Exploratory assessment of cellular immune response to PollenVax | Baseline to Day 50
  Exploratory evaluation of cellular immune response based on changes in Th1/Th2 cytokine profiles in peripheral blood mononuclear cell cultures stimulated with recombinant Art v 1 before and after allergen-specific immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tair Nurpeissov, Principal Investigator — Limited Liability Partnership "Medcenter-Rakhat"
Locations (1):
- Limited Liability Partnership "Medcenter-Rakhat", Almaty, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in publications, including demographic characteristics, safety outcomes (adverse events and serious adverse events), and immunogenicity endpoints (allergen-specific IgE and IgG4 measurements). Data will be fully anonymized and will not include any information that could identify individual participants.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD and supporting documents will be available beginning 6 months after publication of the primary study results and will remain available for up to 5 years thereafter.
Access Criteria: Access to de-identified IPD and supporting documents will be provided to qualified researchers upon reasonable request. Requests must include a research proposal and will be reviewed by the study sponsor and principal investigator. Data will be shared for scientific research purposes only and under a data use agreement that ensures protection of participant confidentiality and intellectual property.

REFERENCES:
- [Result] Tabynov K, Tailakova E, Rakhmatullayeva G, Bolatbekov T, Lim YH, Fomin G, Babayeva M, Valenta R, Tabynov K. Comparison of rArt v 1-based sublingual and subcutaneous immunotherapy in a murine model of asthma. NPJ Vaccines. 2025 Apr 2;10(1):66. doi: 10.1038/s41541-025-01112-1. PMID 40175385